CLINICAL TRIAL: NCT04604041
Title: Investigation of Subclinical Markers of Multiple Sclerosis
Acronym: SUBCLIN-MS
Status: Recruiting | Type: Observational
Sponsor: University of Split, School of Medicine (Other)
Collaborators: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Maja Rogić Vidaković, Research Associate Maja Rogić Vidaković, University of Split, School of Medicine
Other Study IDs: 2181-198-03-04-20-0028.../0005; 003-08/20-03/0005 (Other: University of Split School of Medicine); 2181-147-01/06/M.S.-20-2. (Other: University Hospital of Split); 500-03/20-01/06 (Other: University Hospital of Split)
Record Dates: First submitted 2020-10-02; First posted 2020-10-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis
Keywords: multiple sclerosis; relapsing remitting; TMS; Cytometry; ELISA; corticosteroids; immunomodulation
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum of study participants will be banked for future possible retrospective analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Relapsing-remmitting MS group treated with corticosteroids: 1. Clinical testing
  2. Neurophysiological examination (TMS, EMNG)
  3. Psychomotor examination
  4. Neuropsychological evaluation
  5. Flow cytometry
  6. ELISA
  Interventions: Diagnostic Test: 1. Clinical testing; 2. Neurophysiological examination (TMS, EMNG); 3. Psychomotor examination; 4. Neuropsychological evaluation; 5. Flow cytometry; 6. ELISA
- Relapsing-remmitting MS group treated with immunomodulation: 1. Clinical testing 2. Neurophysiological examination (TMS, EMNG) 4. Neuropsychological evaluation 5. Flow cytometry
  Interventions: Diagnostic Test: 1. Clinical testing; 2. Neurophysiological examination (TMS, EMNG); 3. Psychomotor examination; 4. Neuropsychological evaluation; 5. Flow cytometry; 6. ELISA
- Healthy control group: 5. Flow cytometry
  Interventions: Diagnostic Test: 1. Clinical testing; 2. Neurophysiological examination (TMS, EMNG); 3. Psychomotor examination; 4. Neuropsychological evaluation; 5. Flow cytometry; 6. ELISA

INTERVENTIONS:
Diagnostic Test: 1. Clinical testing; 2. Neurophysiological examination (TMS, EMNG); 3. Psychomotor examination; 4. Neuropsychological evaluation; 5. Flow cytometry; 6. ELISA — All groups will not have the same intervention. Interventions are listed and numbered for each group.

SUMMARY:
Transcranial magnetic stimulation (TMS) studies reported consistent and substantial impairments in the central nervous system (CNS) in multiple sclerosis (MS). Studies of peripheral nervous system (PNS) function comprising electromyoneurography (EMNG) reported impairments of the PNS in MS that were less pronounced and inconsistent. Neurophysiological studies are generally small and cross-sectional and with the poor grouping of MS patients according to MS type.

The objective of the study is to investigate clinical, neurophysiological, and immunological markers in relapsing-remitting MS patients, and in patients with relapsing-remitting MS treated with immunomodulation. The results of the study may contribute to a better understanding of the pathophysiology of multiple sclerosis and can provide guidance in the diagnosis and treatment of patients with relapsing-remitting MS.

DETAILED DESCRIPTION:
The following techniques will be applied:

* Neurophysiological testing will be performed with navigated transcranial magnetic stimulation (nTMS) incorporating an individual MRI of each subject's brain performed on a 1,5 MRI scanner using a series of neuropsychological protocols. Mapping of the primary motor cortex for upper and lower extremity muscles with a recording of motor evoked potentials (MEP) will be performed.
* Electromyoneurography (EMNG) assessment of lower and upper extremities for motor and sensory nerves;
* Neuropsychological assessment will include the general questionnaire and battery of cognitive and psychological tests;
* Immunoassays on blood samples include determination of different markers on monocytes and lymphocytes using flow cytometry, as well as determination of CD163 in serum samples using ELISA.
* Clinical examinations include neurological, biochemical, neuroradiological, and neuropsychological testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a documented diagnosis of relapsing-remitting MS according to the Mc Donald criteria (2005) and with EDSS achievement of 0-3.5 according to the modified Kurtzke's EDSS (Expanded disability status scale) for the assessment of neurological function and incapacity of patients with multiple sclerosis

Exclusion Criteria:

* Patients with metals in the body (e.g. pacemaker, dentures)
* Patients with new pregnancies (verbally confirmed)
* Patients with new head trauma
* Subjects unwilling to sign a consent or follow study procedures

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with documented diagnosis of relapsing-remitting MS according to the McDonald criteria:
  Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Thompson AJ, et al. Lancet Neurol. 2018;17(2):162. Epub 2017 Dec 21
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
TMS assessment of resting motor threshold (RMT) change | RMT before and 5 weeks after steroid intake in relapsing-remitting MS patients. RMT in relapsing-remitting MS group on immunomodulation.
  Neurophysiologic measure of RMT (expressed in percentage of maximal stimulator output) will be evaluated with navigated TMS over the primary motor cortex:
  * in relapsing-remitting MS receiving corticosteroid treatment patients in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
  * relapsing-remitting MS receiving immunomodulation treatment patients at baseline
TMS assessment of motor evoked potentials (MEP) changes from upper and lower extremity muscles | MEP (amplitude and latency) before and 5 weeks after steroid intake in relapsing-remitting MS patients. MEP (amplitude and latency) in relapsing-remitting MS group on immunomodulation.
  The neurophysiologic measure of MEP (amplitude expressed in microvolts and latency expressed in milliseconds) will be evaluated with navigated TMS over the primary motor cortex for upper and lower extremity muscles:
  * in relapsing-remitting MS receiving corticosteroid treatment patients in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
  * relapsing-remitting MS receiving immunomodulation treatment patients at baseline
TMS assessment of cortical silent period (CSP) change | Baseline CSP, CSP change at 5 weeks taking the steroids
  The neurophysiologic measure of CSP duration (expressed in milliseconds) will be evaluated with navigated TMS over the primary motor cortex in relapsing-remitting MS patients in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
TMS assessment of short afferent latency inhibition (SAI) change | Baseline SAI, SAI change at 5 weeks after taking the steroids.
  The neurophysiologic measure of SAI phenomena (expressed in milliseconds) will be evaluated with navigated TMS over the primary motor cortex with peripheral electrical stimulation over the median nerve at different interstimulus intervals (20-28 ms) in relapsing-remitting MS patients in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
EMNG assessment of distal motor latency (DML) and sensory nerve action potential latency (SNAP) change | DML and SNAP latency before and 5 weeks after steroid intake in relapsing-remitting MS patients. DML and SNAP latency in relapsing-remitting MS group on immunomodulation.
  * EMNG measures of DML and SNAP latency (expressed in milliseconds) of upper and lower extremities will be evaluated in relapsing-remitting MS patients receiving corticosteroid treatment in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
  * EMNG measures of DML and SNAP latency (expressed in milliseconds) of upper and lower extremities will be evaluated in relapsing-remitting MS receiving immunomodulation treatment patients at baseline.
EMNG assessment of muscle action potential amplitude (CMAP) and sensory nerve action potential amplitude (SNAP) change | CMAP and SNAP amplitude before and 5 weeks after steroid intake in relapsing-remitting MS patients. CMAP and SNAP amplitude in relapsing-remitting MS group on immunomodulation.
  * EMNG measures of CMAP and SNAP amplitude (expressed in millivolts) of upper and lower extremities will be evaluated in relapsing-remitting MS patients receiving corticosteroid treatment in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
  * EMNG measures of CMAP and SNAP amplitude (expressed in millivolts) of upper and lower extremities will be evaluated in relapsing-remitting MS patients receiving immunomodulation treatment at baseline.
EMNG assessment of motor and sensory conduction velocity (CV) change | CV before and 5 weeks after steroid intake in relapsing-remitting MS patients. CV in relapsing-remitting MS group on immunomodulation.
  * EMNG measures of CV (expressed in meters per second) of motor and sensory nerves of upper and lower extremities will be evaluated in relapsing-remitting MS patients treated with corticosteroids in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
  * EMNG measures of CV (expressed in meters per second) of motor and sensory nerves of upper and lower extremities will be evaluated in relapsing-remitting MS patients treated with immunomodulation treatment at baseline.
EMNG assessment of F-wave change | F-wave before and 5 weeks after steroid intake in relapsing-remitting MS patients. F-wave in relapsing-remitting MS group on immunomodulation.
  -EMNG measures of F-wave (expressed in milliseconds) for motor nerves of upper and lower extremities will be evaluated in relapsing-remitting MS patients treated with corticosteroids in 2 phases (before the intake of steroids, 5 weeks after taking the steroids).
  --EMNG measures of F-wave (expressed in milliseconds) for motor nerves of upper and lower extremities will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline.
CD 14 expression on peripheral blood monocytes change | CD 14 before and 5 weeks after steroid intake in relapsing-remitting MS patients. CD14 in relapsing-remitting MS group on immunomodulation and healthy control group.
  * CD 14 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with corticosteroids in 2 phases (before the intake of steroids, 5 weeks after taking the steroids). The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 14 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline.The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 14 expression on monocytes will be evaluated in the healthy control group.The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
CD 16 expression on peripheral blood monocytes change | CD 16 before and 5 weeks after steroid intake in relapsing-remitting MS patients. CD16 in relapsing-remitting MS group on immunomodulation and healthy control group.
  * CD 16 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with corticosteroids in 2 phases (before the intake of steroids, 5 weeks after taking the steroids). The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 16 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 16 expression on monocytes will be evaluated in the healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
CD 40 expression on peripheral blood monocytes change | CD 40 before and 5 weeks after steroid intake in relapsing-remitting MS patients. CD 40 in relapsing-remitting MS group on immunomodulation and healthy control group.
  * CD 40 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with corticosteroids in 2 phases (before the intake of steroids, and 5 weeks after taking the steroids). The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 40 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 40 expression on monocytes will be evaluated in the healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
CD 192 expression on peripheral blood monocytes change | CD 192 before and 5 weeks after steroid intake in relapsing-remitting MS patients. CD 192 in relapsing-remitting MS group on immunomodulation and healthy control group.
  * CD 192 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with corticosteroids in 2 phases (before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids). The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 192 expression on monocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes.
  * CD 192 expression on monocytes will be evaluated in a healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive monocytes
Change of CD 163 levels in blood serum samples | CD 163 measured before and 5 weeks after taking the steroids.
  CD 163 levels in serum will be evaluated in relapsing-remitting MS patients in 2 phases (before the intake of steroids, 5 weeks after taking the steroids). CD 163 levels will be measured with ELISA assay (expressed in micro mols per litre).
CD 4 expression on lymphocytes | Determination of CD 4 at the beginning of study (study entry) in relapsing-remitting MS patients treated with immunomodulation and in healthy control group.
  * CD 4 expression on lymphocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
  * CD 4 expression on lymphocytes will be evaluated in the healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
CD 25 expression on lymphocytes | Determination of CD 25 at the beginning of study (study entry) in relapsing-remitting MS patients treated with immunomodulation and in healthy control group.
  * CD 25 expression on lymphocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
  * CD 25 expression on lymphocytes will be evaluated in the healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
CTLA-4 expression on lymphocytes | Determination of CTLA-4 at the beginning of study (study entry) in relapsing-remitting MS patients treated with immunomodulation and in healthy control group.
  * CTLA-4 expression on lymphocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
  * CTLA-4 expression on lymphocytes will be evaluated in the healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
FOXP3 expression on lymphocytes | Determination of FOXP3 at the beginning of study (study entry) in relapsing-remitting MS patients treated with immunomodulation and in healthy control group.
  * FOXP3 expression on lymphocytes will be evaluated in relapsing-remitting MS patients treated with immunomodulation at baseline. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
  * FOXP3 expression on lymphocytes will be evaluated in the healthy control group. The expression will be measured as the median of fluorescence distribution acquired with flow cytometry. The expression will also be quantified as the percentage of positive lymphocytes.
Hand dominance assessment with Edinburgh Handedness Inventory test. | Baseline measurement for single subject. The results for all subjects can be provided an average of 1 year of study duration.
  The Edinburgh Handedness Inventory is a well known short questionnaire for determining objectively whether one is left , right handed, or ambidekster. The subjects determines whether he/she is using right or left hand for specific activities (ten activities). The total checks are given for right and left hand, than cumulative sume is given (total checks from right and left hand), difference between total checks for right minus left hand. Final result is the difference result subtracted from cumulative result x 100.
Cognitive assessment change applying Letter Digit Substitution Test (LDST). | Baseline LDST, and LDST change at 5 weeks and 6 months after taking the steroids.
  * Relapsing-remitting MS patients treated with corticosteroids will be tested with LDST before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. LDST is interpreted as the number of correct responses in 60 seconds.
  * Relapsing-remitting MS patients treated with immunomodulation therapy will be tested with LDST at baseline.
Cognitive assessment change applying Montreal Cognitive Assessment (MoCA). | Baseline MoCA, and MoCA change at 5 weeks and 6 months after taking the steroids.
  Relapsing-remitting MS patients will be tested with MoCA before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. MoCA is interpreted as the number of points (30 is maximal).
Psychological assessment change applying Multiple Sclerosis Impact Scale (MSIS-29). | Baseline MSIS-29, and MSIS-29 change at 5 weeks and 6 months after taking the steroids.
  * Relapsing-remitting MS patients treated with corticosteroids will be tested with MSIS before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The total score is formed as the sum of the rounded answers to the two subscales (physical and psychological scale).
  * Relapsing-remitting MS patients treated with immunomodulation will be tested with MSIS at baseline. The total score is formed as the sum of the rounded answers to the two subscales (physical and psychological scale).
Psychological assessment change applying Depression, Anxiety, Stress (DASS-21) scale. | Baseline DASS-21, and DASS-21 change at 5 weeks and 6 months after taking the steroids.
  * Relapsing-remitting MS patients treated with corticosteroids will be tested with DASS-21 before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids.
  * Relapsing-remitting MS patients treated with immunomodulation will be tested with DASS-21 at baseline.
  DASS-21 contains three scales for measuring emotional states of depression, anxiety and stress. Each scale contains 7 statements.
  The result on the depression, anxiety and stress scales is the sum of the rounded answers to specific statements.
Psychological assessment change applying Fatigue Severity Scale (FSS). | Baseline FSS, and FSS change at 5 weeks and 6 months after taking the steroids.
  -Relapsing-remitting MS patients treated with corticosteroids will be tested with FSS before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids.
  --Relapsing-remitting MS patients treated with immunomodulation will be tested with FSS at baseline.
  The subject is asked to read each statement and circle a number from 1 to 7, depending on how appropriate they felt the statement applied to them over the preceding week. A low value indicates that the statement is not very appropriate whereas a high value indicates agreement.The scoring is done by calculating the average response to the questions (adding up all the answers and dividing by nine).
Psychological assessment change applying Pain rating scale. | Baseline Pain rating, and Pain rating change at 5 weeks and 6 months after taking the steroids.
  Relapsing-remitting MS patients will be tested with numerical Pain Rating Scale before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The result is interpreted as the total sum of points. The greater the results the more pain is detected.
Psychomotor assessment of hand grip change applying SAEHAN Squeeze Dynamometer. | Baseline hand grip, and hand grip change at 5 weeks and 6 months after taking the steroids.
  Relapsing-remitting MS patients will be tested with SAEHAN Squeeze Dynamometer before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. Six measurement results are recorded for each subject - three for the grip with the dominant hand and three for the grip with the non-dominant hand. The final result is the mean of the three measurements for each arm expressed in kilograms.
Psychomotor assessment change of extremity muscles applying Lafayette Manual Muscle Tester Dynamometer. | Baseline lower and upper extremity muscle strength, and muscle strength change at 5 weeks and 6 months after taking the steroids.
  Relapsing-remitting MS patients will be tested with Lafayette Manual Muscle Tester Dynamometer before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. Muscle strength measured by Lafayette Manual Muscle Tester is recorded in kilograms and normalized to body-mass index (BMI). Handheld dynamometry will be used to measure ankle dorsiflexion; knee, flexion and extension; hip flexion, extension, abduction, and adduction; and trunk lateral flexion.
Psychomotor assessment change applying Lafayette O'Conner Finger Dexterity Test. | Baseline O'Conner, and O'Conner change at 5 weeks and 6 months after taking the steroids.
  Relapsing-remitting MS patients will be tested with O'Conner Finger Dexterity Test before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The O'Connor Finger Dexterity Test requires hand placement of 3 pins per hole. Result (seconds) = time required to complete the first part of the test + (1.1 x time required to complete the second part of the test) / 2
Barthel Index for Activities of Daily Living (ADL) change. | Baseline activities of daily living, and change in activities of daily living at 5 weeks and 6 months after taking the steroids.
  Relapsing-remitting MS patients will be tested with Barthel Index for Activities of Daily Living (ADL) before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The examiner is rank the patient's independence in the following areas:feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, transfers (bed to chair and back), mobility on level surfaces, and stairs.
  * 0 - 20 = complete dependence; 21 - 60 = severe addiction; 61 - 90 = moderate dependence

SECONDARY OUTCOMES:
-Detection of potential predictors (neurophysiological, neuropsychological, clinical neurological, clinical biochemical, and MRI measures) of medication treatment of relapsing-remitting MS. | The complete data results will be provided at the end of the study.
  Correlation and regression methods will be used to examine the following data:
  * neurophysiological data acquired with TMS (RMT; MEP; CSP; SAI);
  * neurophysiological data acquired with EMNG (DML and SNAP latency; CMAP and SNAP amplitude; motor and sensory CV; F-wave);
  * immunological data (expression profile of CD40, CD192, CD14, CD16 on monocytes and CD25, CTLA-4 and FOXP3 on lymphocytes; expression of CD163 in serum);
  * neuropsychological data; Edinburgh Handedness Inventory test; Pain rating scale; Barthel Index for Activities of Daily Living (ADL); FSS; LDST; MoCA; MSIS-29; DASS-21; O'Conner Finger Dexterity Test; muscle strength - hand grip and upper and lower extremity muscles with a dynamometer
  * clinical: EDSS,T25-FW; MRI; biochemical (complete blood count, differential blood count, AST, ALT, GGT, blood sugar test, creatinine, urine, B12, Na, K, Cl, folic acid, neurotrophic virus in serum and liquor, oligoclonal band)

OTHER OUTCOMES:
Neurological clinical assessment change with Expanded Disability Status Scale (EDSS). | Baseline EDSS, and EDSS change at 5 weeks and 6 months after taking the steroids.
  * EDSS applied in relapsing-remiting MS patients before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids.
  * EDSS applied in relapsing-remiting MS patients treated with immunomodulation at baseline.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Neurological clinical assessment change with Timed 25-Foot Walk (T25-FW). | Baseline T25-FW, and T25-FW change at 5 weeks and 6 months after taking the steroids.
  T25-FW applied in relapsing-remiting MS patients before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids.The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The score for the T25-FW is the average of the two completed trials.
Clinical biochemical assessment change of complete blood count. | Baseline complete blood count, and blood coun change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of differential blood count will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. Following components of the blood are measured: leukocytes (x10^9/L) (ref. interval. 3.4-9.7), erythrocytes (x10^12/L) (ref. interval 3.86-5.08), haemoglobin (g/L) (ref. interval 119-157), hematocrit (L/L) (ref. interval 0.356-0.470), MCV (fL) (ref. interval 83.0-97.2), MCH (pg) (ref. interval 27.4-33.9), MCHC (g/L) (ref. interval 320-345), index of scattering of erythrocytes (%) (ref. interval 9.0-15.0), thrombocytes (x10^9/L) (ref. interval 158-424), MPV (fL) (ref. interval 6.8-10.4), PDW (%) (ref. interval 35-65), PCT (L/L) (ref. interval 0.001-0.004)
Clinical biochemical assessment change of differential blood count. | Baseline differential blood count, and differential blood count change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of differential blood count will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The blood collection is taken early in the morning, before breakfast. Following components of the blood are measured: neutrophile granulocytes (%) ( ref. interval 44-72), lymphocyte (%) (ref. interval 20-46), monocyte (%) (ref.interval 2-12), eosinophile (%) (ref. interval 0-7), basophile (%) (ref. interval 0-1), neutrophile # (x10^9/L) (ref. interval 2.06-6.49), lymphocyte # (x10^9/L) (ref. interval 1.19-3.35), monocyte # (x10^9/L) (ref. interval 0.12-0.84), eosinophile # (x10^9/L) (ref. interval 0.00-0.43), basophile # (x10^9/L) (0.00-0.06)
Clinical biochemical assessment change of glucose. | Baseline glucose, and glucose change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of glucose will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The glucose is measured in mmol/L, and ref. interval is 4.4-6.4
Clinical biochemical assessment change of urea. | Baseline urea, and urea change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of urea will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The urea is measured in mmol/L, and ref. interval is 2.8-8.3
Clinical biochemical assessment change of creatinine. | Baseline creatinine, and creatinine change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of creatinine will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The creatinine is measured in micro mol/L, and ref. interval is 49-90
Clinical biochemical assessment change of Aspartate Aminotransferase (AST) Test. | Baseline AST, and AST change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of AST test will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. A high AST level is a sign of liver damage, but it can also mean the patient have damage to another organ like heart or kidneys. The normal range of values for AST is about 8 to 30 units per liter of serum (the liquid part of the blood).
Clinical biochemical assessment change of Alanine Aminotransferase (ALT) Test. | Baseline ALT, and ALT change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of ALT test will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. A high ALT level is a sign of liver damage, but it can also mean the patient have damage to another organ like heart or kidneys. The normal range of values for ALT is about 10 to 36 units per liter of serum (the liquid part of the blood).
Clinical biochemical assessment change of Gamma-Glutamyl Transferase (GGT). | Baseline GGT, and GGT change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of GGT test will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. GGT is elevated in the blood in most diseases that cause damage to the liver or bile ducts. The normal range for GGT levels is 9-35 units per liter (U/L). Normal values can vary due to age and sex.
Clinical biochemical assessment change of urine. | Baseline urine, urine change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of urine will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. Urine examination will include colour (expressed as a qualitative unit), acidity (pH, ref. interval 5-9), specific gravity (kg/L, 1.002-1.030), glucose (pos or neg), bilirubin (pos or neg), ketones (pos or neg), haemoglobin (pos or neg), proteins (pos or neg), urobilinogen (pos or neg).
Clinical biochemical assessment change of B12. | Baseline B12, B12 change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of B12 will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The normal range for vitamin B12 can vary slightly depending on the lab. But a normal level of vitamin B12 in blood is generally between 145 and 569 picomols per litre (pmol/L).
Clinical biochemical assessment change of sodium (Na). | Baseline Na, Na change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of Na will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The normal range for blood sodium levels is 137 to 146 millimoles per litre (mmol/L).
Clinical biochemical assessment change of potassium (K). | Baseline K, K change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of K will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The normal range for blood potassium levels is 3.9 to 5.1 millimoles per litre (mmol/L).
Clinical biochemical assessment change of chloride (Cl). | Baseline Cl, Cl change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of Cl will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The normal range for Cl levels is 97 to 108 millimoles per litre (mmol/L).
Clinical biochemical assessment change of folic acid (FA). | Baseline FA, and FA change at 5 weeks and 6 months after taking the steroids.
  Clinical biochemical assessment of FA will be provided before the intake of steroids, 5 weeks after taking the steroids and 6 months after taking the steroids. The normal range for FA levels is 8.83 to 60.8 nanomoles per litre (nmol/L).
Serologic test for neurotropic viruses and bacteria in blood serum and cerebrospinal liquor. | Baseline Serologic test for neurotropic viruses and bacteria in blood serum and cerebrospinal liquor.
  Serologic test for neurotropic viruses and bacteria in blood serum and cerebrospinal liquor will be provided before the intake of steroids. Seroconversion for Epstein Barr virus, Cytomegalovirus, Herpes simplex 1/2 virus, Borrelia burgdoferi, German measles virus, Measles virus. Seroconversion is expressed as positive or negative.
Microscopic and biochemical assessment of cerebrospinal liquor. | Baseline Microscopic and biochemical assessment of cerebrospinal liquor
  Microscopic and biochemical assessment of cerebrospinal liquor includes: colour (qualitative units), transparency (qualitative units), leukocytes # (10^6/L), erythrocytes # (10^6/L), glucose (mmol/L, ref interval 2.49 to 4.44), lactate (mmol/L, ref interval 1.1-2.2), total protein (mg/L, ref interval 170-370) , chlorides (mmol/L, ref interval 115-129)
Oligoclonal bands in cerebrospinal liquor. | Baseline Oligoclonal bands in cerebrospinal liquor
  Oligoclonal bands in cerebrospinal liquor will be assessed at baseline, measured as present or absent.
MRI radiological evaluation with contrast for detection of plaques and plaque location. | MRI scanning baseline and 6 months after the intake of steroids.
  * Each MS patient treated with corticosteroid will have MRI scanning before intake of steroids and 6 months after the intake. Number and location of different radiological lesions will be noted.
  * Each MS patient treated with immunomodulation will have MRI scanning at baseline (also verifying pre-baseline MRI if available).

CONTACTS AND LOCATIONS:
Overall Officials: Maja Rogić Vidaković, MSc, PhD, Principal Investigator — University of Split, School of Medicine
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Mamoei S, Hvid LG, Boye Jensen H, Zijdewind I, Stenager E, Dalgas U. Neurophysiological impairments in multiple sclerosis-Central and peripheral motor pathways. Acta Neurol Scand. 2020 Nov;142(5):401-417. doi: 10.1111/ane.13289. Epub 2020 Jun 23. PMID 32474916
- [Background] Gorgulu U, Ergun U, Ertugrul L. Peripheral nerve conductions in relapsing remitting multiple sclerosis (RRMS) patients. J Clin Neurosci. 2020 Apr;74:93-97. doi: 10.1016/j.jocn.2020.01.058. Epub 2020 Feb 3. PMID 32029369
- [Background] Gjelstrup MC, Stilund M, Petersen T, Moller HJ, Petersen EL, Christensen T. Subsets of activated monocytes and markers of inflammation in incipient and progressed multiple sclerosis. Immunol Cell Biol. 2018 Feb;96(2):160-174. doi: 10.1111/imcb.1025. Epub 2017 Dec 11. PMID 29363161
- [Background] Howard LM, Miga AJ, Vanderlugt CL, Dal Canto MC, Laman JD, Noelle RJ, Miller SD. Mechanisms of immunotherapeutic intervention by anti-CD40L (CD154) antibody in an animal model of multiple sclerosis. J Clin Invest. 1999 Jan;103(2):281-90. doi: 10.1172/JCI5388. PMID 9916140
- [Background] Kawarabayashi R, Motoyama K, Nakamura M, Yamazaki Y, Morioka T, Mori K, Fukumoto S, Imanishi Y, Shioi A, Shoji T, Emoto M, Inaba M. The Association between Monocyte Surface CD163 and Insulin Resistance in Patients with Type 2 Diabetes. J Diabetes Res. 2017;2017:6549242. doi: 10.1155/2017/6549242. Epub 2017 Dec 28. PMID 29445750
- [Background] Wojcik CM, Beier M, Costello K, DeLuca J, Feinstein A, Goverover Y, Gudesblatt M, Jaworski M 3rd, Kalb R, Kostich L, LaRocca NG, Rodgers JD, Benedict RH; National MS Society Cognition Work Team. Computerized neuropsychological assessment devices in multiple sclerosis: A systematic review. Mult Scler. 2019 Dec;25(14):1848-1869. doi: 10.1177/1352458519879094. Epub 2019 Oct 22. PMID 31637963
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Result] Jerkovic A, Matijaca M, Prorokovic A, Sikic A, Kosta V, Curkovic Katic A, Dolic K, Duka Glavor K, Soda J, Dogas Z, Rogic Vidakovic M. Information Processing Speed Assessed with Letter Digit Substitution Test in Croatian Sample of Multiple Sclerosis Patients. Diagnostics (Basel). 2022 Jan 4;12(1):111. doi: 10.3390/diagnostics12010111. PMID 35054278
- [Result] Jerkovic A, Prorokovic A, Matijaca M, Vuko J, Poljicanin A, Mastelic A, Curkovic Katic A, Kosta V, Kustura L, Dolic K, Ethogas Z, Rogic Vidakovic M. Psychometric Properties of the HADS Measure of Anxiety and Depression Among Multiple Sclerosis Patients in Croatia. Front Psychol. 2021 Nov 30;12:794353. doi: 10.3389/fpsyg.2021.794353. eCollection 2021. PMID 34917005
- [Result] Rogic Vidakovic M, Simic N, Poljicanin A, Nikolic Ivanisevic M, Ana J, Dogas Z. Psychometric properties of the Croatian version of the depression, anxiety, and stress scale-21 and multiple sclerosis impact scale-29 in multiple sclerosis patients. Mult Scler Relat Disord. 2021 May;50:102850. doi: 10.1016/j.msard.2021.102850. Epub 2021 Feb 20. PMID 33636617
- [Derived] Bralic A, Pavelin S, Pleic N, Soda J, Dolic K, Markotic A, Curkovic Katic A, Mastelic A, Rezic Muzinic N, Duranovic J, Kljajic Z, Stipica Safic I, Dogas Z, Rogic Vidakovic M. Correspondence of MRI and nTMS With EDSS in Multiple Sclerosis: Longitudinal Follow-Up Study. Ann Clin Transl Neurol. 2025 Jun;12(6):1240-1255. doi: 10.1002/acn3.70041. Epub 2025 Apr 17. PMID 40244940